CLINICAL TRIAL: NCT04143269
Title: Treatment of Complications to Diabetic Autonomic Neuropathy With Vagus Nerve Stimulation
Acronym: DAN-VNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Principal Investigator, Asbjørn Mohr Drewes, Professir, Chief Physician, MD, PhD, DMSc, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAN-VNS; CIV-19-07-029105 (Other: Danish Health and Medicines Authority); N-20190020 (Other: North Denmark Region Committee in Health Research Ethics)
Record Dates: First submitted 2019-10-22; First posted 2019-10-29 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Gastrointestinal Dysfunction; Diabetes Mellitus
Keywords: Vagal nerve stimulation; Gastrointestinal symptoms; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active treatment (Active Comparator): Non-invasive transcutaneous vagus nerve stimulation applied by the GammaCore device (ElectroCore LLC)
  Interventions: Device: Non-invasive transcutaneous vagus nerve stimulation
- Sham Treatment (Sham Comparator): Inactive sham vagus nerve stimulation applied by the GammaCore sham device (ElectroCore LLC)
  Interventions: Device: Sham vagus nerve stimulation

INTERVENTIONS:
Device: Non-invasive transcutaneous vagus nerve stimulation — Bilateral stimulation 4 times per day for 7 days (period 1) and 2 times per day for 8 weeks (period 2). The two periods are separated by a 2 weeks wash-out period.
  Other Names: GammaCore device
  Arms: Active treatment
Device: Sham vagus nerve stimulation — Bilateral stimulation 4 times per day for 7 days (period 1) and 2 times per day for 8 weeks (period 2). The two periods are separated by a 2 weeks wash-out period.
  The sham device produces a slight vibrating sensation, but do not provide any vagal nerve activation
  Other Names: GammaCore sham device
  Arms: Sham Treatment

SUMMARY:
The purpose of the DAN-VNS study is to investigate the effects of non-invasive vagal nerve stimulation on gastrointestinal symptoms such as nausea, vomiting, bloating, and diarrhea in people with diabetes.

DETAILED DESCRIPTION:
The study is a randomized, double-blinded, sham-controlled, parallel group clinical trial, which will include participants with diabetes and gastrointestinal (GI) problems. These problems may be manifestations of diabetic autonomic neuropathy.

Participants are randomised to received either active non-invasive transcutaneous vagal nerve stimulation (tVNS) or inactive sham stimulation. The study period is divided in two phases. The first phase investigates the effects of short-term, high-intensity tVNS treatment on GI symptoms. The second phase investigates the effects of long-term, middle-intensity tVNS treatment. The primary outcome of both phases is subjective patient evaluation of GI symptoms by the use of validated questionnaires.

A third phase, conducted only on participants, who proved to be responsive to tVNS treatment, will investigate the acute endocrine and metabolic response to short-term tVNS in a randomised cross-over design.

Lastly, healthy volunteers will be included in a cross-sectional, descriptive study in order to provide a comparable baseline dataset.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Verified diagnosis of diabetes for a minimum of 1 year and with stable medication
* CAN-score ≥ 1 (measured by the Vagus device (Medicus Engineering, Aarhus, Denmark) OR COMPASS-31 score of ≥ 16 OR electrochemical resistance <50µS (hands) and <70µS (feet) assessed with the SUDOSCAN device
* Weighted composite score of Gastroparesis Cardinal Symptom Index (GCSI) and Gastrointestinal Symptom Rating Scale (GSRS) ≥ 2.3
* Ability to read and understand Danish
* Personally signed and dated informed consent documents
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures

Exclusion Criteria:

* Significant GI diseases not related to diabetes
* Significant cardiovascular diseases
* GI surgery within 3 months prior to study inclusion
* Swallowing disorders
* Blood pressure < 100/60 or > 160/105
* Clinically significant bradycardia or tachycardia
* Implanted portable electro-mechanical medical devices including pacemaker, defibrillator, cochlear implant, and infusion pump
* Previous surgery of the vagus nerve
* Active laser treatment for proliferative retinopathy
* Contraindications for MRI
* Any clinical abnormalities, that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results
* Pregnancy or intention to become pregnant or father a child during the course of the study
* Participation in other clinical trials less than three months prior to inclusion, unless such a participation is judged to have no influence on the recordings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Subjective gastrointestinal symptoms | At baseline and after 7 days (period 1) and 8 weeks (period 2) of intervention
  Assessed as changes from baseline in scores from the validated questionnaire Gastroparesis Cardinal Symptom Index (GCSI). The GCSI-score ranges from 0 to 5 with a higher score indicating a higher amount of experienced symptoms
Subjective gastrointestinal symptoms | At baseline and after 7 days (period 1) and 8 weeks (period 2) of intervention
  Assessed as changes from baseline in scores from the validated questionnaire Gastrointestinal Symptom Rating Scale (GSRS). The GSRS-score ranges from 1 to 7 with a higher score indicating a higher amount of experienced symptoms

SECONDARY OUTCOMES:
Holter monitoring | At baseline and after 7 days (period 1) of intervention
  A small patch sensor (ePatch) will be used to monitor the heart rate variability during a period of 5 days. Classical time (RR-interval, SDNN, SDNNi, SDANN, RMSSD) and frequency (VLF, LF, HF and LF/HF) domain heart rate variability parameters will be assessed
Cardiac vagal tone | At baseline and after 7 days (period 1) of intervention
  A three lead electrocardiography device (eMotion Faros) will record the cardiac vagal tone during a period of 5 minutes rest. Cardiac vagal tone is measured on a linear vagal scale with a low score indicating dysfunction of the vagal nerve
Cardiovascular reflex testing | At baseline and after 7 days (period 1) of intervention
  The VAGUS device, will be used to test three different standardised heart reflexes(Ewings battery). From these tests the device calculates a score from 0-3 indicating the degree of autonomic neuropathy, with 0 being no neuropathy and 3 being manifest neuropathy
Sudomotor function | At baseline and after 7 days (period 1) of intervention
  Measured by SUDOSCAN device
Pan-intestinal imaging | At baseline and after 7 days (period 1) of intervention
  By MR scanning
Functional brain scan | At baseline and after 7 days (period 1) of intervention
  By MR scanning
Intestinal transit | At baseline and after 8 weeks (period 2) of intervention
  Participants will swallow a indigestible wireless motility capsule (SmartPill) in order to assess the transit time of whole gut as well as individual segments.
EEG spectral analysis | At baseline and after 7 days (period 1) of intervention
  40 electrodes will be used to record EEG during a period of 5 minutes rest. The results will be used to model connectivity between brain centres as well as the dominating centres of brain. EEG power will be assessed in the Delta, Theta, Alpha, Beta, and Gamma bands between 1 and 70 Hertz. Finally inverse modelling will be conducted to explore the dominating centres of brain activity.
Pain tolerance threshold | At baseline and after 7 days (period 1) of intervention
  Pressure will be applied to the tibial bone and the quadriceps muscle by a handheld pressure algometer. The pain tolerance threshold (measured in kPa) is reached when the participant reports the pain to be intolerable
Cold pressor test | At baseline and after 7 days (period 1) of intervention
  The left hand of the participant is immersed in 2.0 degree (celsius) cold water for up to 2 minutes or until the pain becomes intolerable. The participant is asked to rate the pain on a 10-point Visual Analogue Scale (0 being no pain and 10 being worst imaginable pain) every 10 seconds during the test.
Glycaemic control | At baseline and after 7 days (period 1) and 8 weeks (period 2) of intervention
  Continuous glucose monitoring (FreeStyle Libre)
Level of inflammation | At baseline and after 7 days (period 1) and 8 weeks (period 2) of intervention
  Multiplex analysis of serum samples. Serum concentrations (pg/mL) of inflammatory biomarkers (TNF-alpha, IL-2, IL-4, IL-6 and IL-10) will be assessed.
24-hours blood pressure | At baseline and 8 weeks (period 2) of intervention
  Participants wear a device for 24 hours, whivh measures blood pressure (systolic and diastolic) every 15 minutes during daytime and every 30 minutes during the night
Kidney function | At baseline and 7 days (period 1) and 8 weeks (period 2) of intervention
  Participants deliver morning urine samples and urine albumine and urin creatinine will be measured.
Nerve conduction study - velocities | At baseline in period 1
  Nerve conduction test of large fibre function will be performed. Velocities of motor and sensory nerves (peroneal, tibial, ulnar, sural, radial, and median) will be assesed.
Nerve conduction study - amplitudes | At baseline in period 1
  Nerve conduction test of large fibre function will be performed. Amplitudes of motor and sensory nerves (peroneal, tibial, ulnar, sural, radial, and median) will be assesed.

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, Professor, Principal Investigator — Aalborg University Hospital
Locations (1):
- Steno Diabetes Center North Jutland, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can be provided upon request.
Time Frame: From study end. No end date
Access Criteria: Researchers who provide a methodological sound proposal

REFERENCES:
- [Derived] Kornum DS, Bertoli D, Kufaishi H, Wegeberg AM, Okdahl T, Mark EB, Hoyer KL, Frokjaer JB, Brock B, Krogh K, Hansen CS, Knop FK, Brock C, Drewes AM. Transcutaneous vagal nerve stimulation for treating gastrointestinal symptoms in individuals with diabetes: a randomised, double-blind, sham-controlled, multicentre trial. Diabetologia. 2024 Jun;67(6):1122-1137. doi: 10.1007/s00125-024-06129-0. Epub 2024 Mar 28. PMID 38546822
- [Derived] Okdahl T, Bertoli D, Brock B, Krogh K, Knop FK, Brock C, Drewes AM. Study protocol for a multicentre, randomised, parallel group, sham-controlled clinical trial investigating the effect of transcutaneous vagal nerve stimulation on gastrointestinal symptoms in people with diabetes complicated with diabetic autonomic neuropathy: the DAN-VNS Study. BMJ Open. 2021 Jan 6;11(1):e038677. doi: 10.1136/bmjopen-2020-038677. PMID 33408197